CLINICAL TRIAL: NCT02086591
Title: A Phase II Study of Doxycycline in Relapsed NHL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Carla Casulo, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50370; 120145 (Other: IND)
Record Dates: First submitted 2014-02-26; First posted 2014-03-13 (Estimated); Results first posted 2016-12-22 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-10

CONDITIONS: Adult Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma Recurrent; Lymphoma, Follicular; Marginal Zone B-Cell Lymphoma; Malignant Lymphoma - Lymphoplasmacytic; Waldenstrom Macroglobulinemia; Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia (CLL); T-Cell Lymphoma
Keywords: Non Hodgkin Lymphoma; Doxycycline
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, T-Cell; Lymphoma, Non-Hodgkin | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxycycline (Experimental): Doxycycline 200 mg twice daily
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline

SUMMARY:
The purpose of this study is to determine whether doxycycline is effective in the treatment of relapsed Non Hodgkin Lymphomas (NHL).

DETAILED DESCRIPTION:
The long-term objective of this proposal is to develop more effective and less toxic therapeutic approaches for relapsed and refractory Non Hodgkin Lymphomas (NHL). Given the incurability of indolent lymphomas, innovative strategies for treatment are needed. For aggressive lymphomas such as Diffuse Large B Cell Lymphoma (DLBCL), novel treatments are particularly relevant since one third of patients have disease that will relapse or is refractory to standard therapy. Outcomes for this remaining group of patients are very poor. To address this unmet need, we have identified the antimicrobial agent doxycycline as a novel drug repurposed for lymphoma treatment based on results from a small molecule screen against Diffuse Large B Cell Lymphoma (DLBCL). Through preclinical work in his laboratory, my basic science collaborator Dr. Jiyong Zhao has found that doxycycline inhibits proliferation and survival in both activated B cell (ABC) type and germinal center B (GCB) type Diffuse Large B Cell Lymphoma (DLBCL) cell lines, as well as in Burkitt lymphoma (BL) and follicular lymphoma (FL) cell lines. Based on this preliminary data, we propose an open label, single center phase II study of doxycycline in patients with relapsed Non Hodgkin Lymphomas (NHL). We have selected a dose and schedule (200 mg BID by mouth daily) based on maximum antimicrobial dose use, and acceptance of tolerability in several studies. The planned correlative studies should help to identify potential biomarkers for response to doxycycline, such as plasma matrix metalloproteinase 9 (MMP9), and provide further insight into potential mechanisms of doxycyline action hypothesized from results of prior laboratory studies.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed aggressive or indolent NHL following any prior treatment of the following etiologies:

  * Diffuse large B cell lymphoma (DLBCL)
  * Mantle cell lymphoma (MCL)
  * Follicular lymphoma (FL)
  * Marginal zone lymphoma (MZL)
  * Lymphoplasmacytic lymphoma (LPL)
  * Waldenstrom's macroglobulinemia (WM)
  * Small lymphocytic lymphoma (SLL)
  * Chronic lymphocytic leukemia (CLL)
  * T cell lymphoma (TCL)
* Ages ≥ 18
* Karnofsky Performance Status (KPS) ≥ 60% or Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤2
* Life expectancy of at least 3 months
* Measurable disease in at least one target lesion, assessable by radiographic examination with Fludeoxyglucose-Positron Emission Tomography (FDG-PET) or computed tomography (CT), bone marrow evaluation showing involvement, or peripheral blood showing involvement of lymphoma
* Adequate organ function:

  * Absolute neutrophil count (ANC) > 500 cells/mL and platelet count > 50,000 cells/mL unless felt to be secondary to lymphoma at which any count is permissible.
  * Adequate renal function as determined by Creatinine (Cr) < 1.5x upper limit of normal (ULN) or estimated creatinine clearance of ≥ 60mL/min
  * Adequate hepatic function as determined by total bilirubin < 1.5x upper limit of normal (ULN) (unless known Gilbert syndrome), alanine aminotransferase (ALT)and aspartate aminotransferase (AST) < 2.5x upper limit of normal (ULN)

Exclusion Criteria:

* Known sensitivity or allergy to tetracyclines
* Lack of measurable disease by computed tomography (CT) or Fludeoxyglucose-Positron Emission Tomography (FDG-PET)
* Karnofsky Performance Status (KPS) <60% or Eastern Cooperative Oncology Group Performance Status (ECOG PS) >2
* Curative treatment is indicated or possible
* Inadequate organ function as measured by not fulfilling above criteria
* Pregnancy, positive serum human chorionic gonadotropin (hCG) within 28 days of enrollment, or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-03; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Casulo, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Doxycycline: Doxycycline 200 mg twice daily
  Doxycycline
Period: Overall Study
Arm/Group | Doxycycline
Started | 7
Completed | 2
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — protocol terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Doxycycline
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Gender [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of patients with disease progression. Progression is defined as:
  * Appearance of a new lesion on fluorodeoxyglucose (FDG)-positron emission tomography or computerized tomography
  * ≥50% increase in sum of the product of the node dimensions (SPD) of more than one node or in greatest diameter of any previously identified node >1 cm in its short axis from nadir.
  * To be considered progressive disease, a lymph node with a diameter of the short axis of less than 1.0 cm must increase by 50% and to a size of 1.5 x 1.5 cm or more than 1.5 cm in the long axis.
  * At least a 50% increase in the longest diameter of any single previously identified node more than 1 cm in its short axis.
Time Frame: Three months
Measure: Number; unit: percentage of participants
Arm/Group | Doxycycline
Number analyzed (Participants) | 7
percentage of participants | 28

2. Secondary Outcome: Percentage of Patients With Progression Free Survival
Description: Progression free survival is defined as the percentage of patients with stable disease or no death. Stable disease is defined as less than a partial response but is not progressive disease. Partial Response (PR)-At least a 50% decrease in sum of the product of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses as determined byFDG-PET for CT scan. No increase should be observed in the size of other nodes, liver, or spleen. Patients who achieve a CR by the above criteria, but who have persistent morphologic bone marrow involvement will be considered partial responders. When the bone marrow was involved before therapy and a clinical CR was achieved, but with no bone marrow assessment after treatment, patients should be considered partial responders.
Time Frame: One year
Population: Data was collected on all patients who were enrolled.
Measure: Number; unit: percentage of participants
Arm/Group | Doxycycline
Number analyzed (Participants) | 7
percentage of participants | 57

3. Other Pre Specified Outcome: Exploratory Objective
Description: To investigate change in plasma matrix metalloproteinase 9 (MMP9) levels as a biomarker of treatment response; to assess plasma matrix metalloproteinase 9 (MMP9) expression by immunohistochemistry (IHC) and correlate to response in order to test the hypothesis that elevated intratumoral levels of plasma matrix metalloproteinase 9 (MMP9) can predict response to doxycycline. To assess activation/expression of nuclear factor kappa-light-chain-enhancer of activated B cells (NF-kb) and Signal transducer and activator of transcription 3 (STAT 3) pathways in archived tumor by immunohistochemistry (IHC) to predict response or resistance to doxycycline.
Time Frame: One year
Population: No data displayed because Outcome Measure has zero total participants analyzed
Arm/Group | Doxycycline
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Doxycycline
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Doxycycline (N=7)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3
musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1
alanine aminotransferase increase (Investigations) | 1
creatinine increased (Investigations) | 1
sepsis (Infections and infestations) | 1
vomiting (Gastrointestinal disorders) | 2
nausea (Gastrointestinal disorders) | 6
fatigue (General disorders) | 2
face edema (General disorders) | 1
pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes